CLINICAL TRIAL: NCT04253626
Title: Comparison of Oral Ferrous Sulfate to Intravenous Ferumoxytol in Antepartum Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Deirdre Lyell, Professor, Obstetrics & Gynecology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 54788; K12HD103084 (NIH)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related; Anemia, Iron Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous iron (Experimental): Participants will receive 510mg intravenous iron ferumoxytol, with a maximum of 2 doses based on the baseline hemoglobin level. The ferumoxytol is administered as an infusion for approximately 15 - 30 minutes.
  Interventions: Drug: Ferumoxytol Injection [Feraheme]
- Oral iron (Active Comparator): Participants will be prescribed 1-2 ferrous sulfate 325mg tablets by mouth (based on severity of anemia) until delivery. For standardization, the dosage is as follows based on severity: one ferrous sulfate tablet for women with baseline hemoglobin 9-11, and two ferrous sulfate tablets for hemoglobin < 9.
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Ferumoxytol Injection [Feraheme] — 510mg intravenous ferumoxytol
  Arms: Intravenous iron
Drug: Ferrous Sulfate — 325mg oral ferrous sulfate
  Arms: Oral iron

SUMMARY:
Evaluate the extent to which treatment of iron deficiency anemia beyond 24-34 weeks' gestation of pregnancy with intravenous iron increases hemoglobin compared to oral iron. The investigators will test the hypothesis that pregnant women who are anemic in the second and third trimester are more likely to significantly increase their hemoglobin with intravenous iron as opposed to the usual standard of care, oral iron.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women 18 years old and above
2. Hemoglobin < 11 g/dL, serum ferritin < 30 ug/dL and or transferrin saturation (TSAT) < 20%
3. Between 24-34 weeks' pregnancy
4. Singleton pregnancy
5. Receiving prenatal care at Stanford/LPCH OB clinic and planning to deliver at LPCH
6. Hemodynamically stable

Exclusion Criteria:

1. Patients unable to give informed consent
2. Known allergy/hypersensitivity to IV iron
3. Inflammatory Bowel Disease or history of gastric bypass surgery
4. Dialysis-dependent Chronic Kidney Disease/ ESRD
5. Known Hemoglobinopathies such as sickle cell disease, beta-thalassemia, alpha thalassemia
6. Folate/Vitamin B12 deficiency
7. Known malignancy
8. Medication allergy to Tylenol (acetaminophen)
9. Hemoglobin above 12 or less than 7 g/dL
10. Patients with complex past medical histories which may include history of multiple medication allergies (greater than 2 allergies), connective tissue disorder, etc.
11. Diagnosis of placenta previa

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Lyell, Principal Investigator — Stanford University; Irogue Igbinosa, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine/Lucile Packard Childrens Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Can describe study design here, up to 500 characters with spaces
Pre-assignment Details: 83 participants signed informed consent; 80 were allocated to treatment.
Groups:
- Oral Iron: Participants are prescribed 1-2 ferrous sulfate 325mg tablets by mouth (based on severity of anemia) until delivery.
- Intravenous Iron: Participants receive 510mg intravenous iron ferumoxytol, with a maximum of 2 doses based on the baseline hemoglobin level.
Period: Overall Study
Arm/Group | Oral Iron | Intravenous Iron
Started | 40 | 40
Received Allocated Intervention | 39 | 38
Discontinued Intervention | 6 | 1
Analyzed for Primary Outcome | 38 | 36
Completed | 38 | 36
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Population: Intention to treat; all participants were analyzed according to the group to which they were randomized, regardless of treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Iron | Intravenous Iron | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.0 [30.8 to 35.5] | 32.0 [29.0 to 35.0] | 32.0 [29.0 to 35.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latine | 11 | 11 | 22
  Non Hispanic Asian or Pacific Islander | 11 | 12 | 23
  Non Hispanic Black or African American | 2 | 4 | 6
  Non Hispanic White | 12 | 12 | 24
  Other/Unknown | 4 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Median Change in Hemoglobin Value Before and After Intervention
Description: Hemoglobin is measured as g/dL at enrollment and after the study intervention
Time Frame: From enrollment to four weeks post-enrollment (may have been up to 6 weeks post-enrollment)
Population: Participants analyzable for the primary outcome (had data through week 4)
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Oral Iron | Intravenous Iron
Number analyzed (Participants) | 38 | 36
g/dL | 10.95 [9.88 to 11.18] | 11.45 [11.13 to 12.03]
Statistical Analysis 1: Comparison: Oral Iron vs Intravenous Iron; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05

2. Secondary Outcome: Number of Participants Who Discontinued Treatment
Time Frame: From enrollment to delivery or birth admission (average approximately 8 to 12 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Iron | Intravenous Iron
Number analyzed (Participants) | 40 | 40
Participants | 6 | 1

3. Secondary Outcome: Number of Participants With Serious Adverse Events Associated With Treatment
Time Frame: From enrollment to delivery or birth admission (average approximately 8 to 12 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Iron | Intravenous Iron
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

4. Secondary Outcome: Number of Participants Who Need Blood Transfusion Postpartum
Time Frame: From enrollment to delivery or birth admission (average approximately 8 to 12 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Iron | Intravenous Iron
Number analyzed (Participants) | 40 | 40
Participants | 3 | 0

5. Secondary Outcome: Change in Short Form (SF-)36 General Health Symptom Score
Description: Score range: 0 to 100 (lower scores indicate more severe symptoms, higher scores correspond to fewer symptoms)
Time Frame: From enrollment to four weeks post-enrollment (may have been up to 6 weeks post-enrollment)
Population: Participants with data at the respective time point
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Oral Iron | Intravenous Iron
Number analyzed (Participants) | 39 | 38
score on a scale
  Baseline | 63 [44 to 63] | 63 [50 to 63]
  Change at week 4: number analyzed (Participants) | 36 | 34
  Change at week 4 | 0 [-13 to 3] | 0 [-13 to 0]
Statistical Analysis 1: Comparison: Oral Iron vs Intravenous Iron; Between-group analysis of change at week 4; Test type: Other; p = 0.88, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was < 0.05

6. Secondary Outcome: Change in Short Form (SF-)36 Physical Functioning Score
Description: Score range: 0 to 100 (lower scores indicate less physical function, higher scores correspond to more physical function).
Time Frame: From enrollment to four weeks post-enrollment (may have been up to 6 weeks post-enrollment)
Population: Participants with data at the respective time point
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Oral Iron | Intravenous Iron
Number analyzed (Participants) | 39 | 38
score on a scale
  Baseline | 70 [65 to 80] | 70 [50 to 90]
  Change at week 4: number analyzed (Participants) | 35 | 34
  Change at week 4 | -10 [-20 to 5] | 0 [-18 to 10]
Statistical Analysis 1: Comparison: Oral Iron vs Intravenous Iron; Between-group analysis of change at week 4; Test type: Other; p = 0.27, Wilcoxon (Mann-Whitney); The a priori threshold for statistical significance was < 0.05

7. Secondary Outcome: Change in Short Form (SF-)36 Role Limitations Due to Physical Health Score
Description: Score range: 0 to 100 (lower scores indicate more limitations, higher scores correspond to fewer limitations).
Time Frame: From enrollment to four weeks post-enrollment (may have been up to 6 weeks post-enrollment)
Population: Participants with data at the respective time point
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Oral Iron | Intravenous Iron
Number analyzed (Participants) | 38 | 37
score on a scale
  Baseline | 38 [0 to 100] | 50 [0 to 100]
  Change at week 4: number analyzed (Participants) | 33 | 36
  Change at week 4 | 0 [0 to 25] | 0 [0 to 50]
Statistical Analysis 1: Comparison: Oral Iron vs Intravenous Iron; Between-group analysis of change at week 4; Test type: Other; p = 0.72, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was < 0.05

8. Secondary Outcome: Change in Short Form (SF-)36 Energy/Fatigue Score
Description: Score range: 0 to 100 (lower scores indicate more fatigue, higher scores correspond to more energy).
Time Frame: From enrollment to four weeks post-enrollment (may have been up to 6 weeks post-enrollment)
Population: Participants with data at the respective time point
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Oral Iron | Intravenous Iron
Number analyzed (Participants) | 39 | 38
score on a scale
  Baseline | 50 [30 to 60] | 40 [23 to 60]
  Change at week 4: number analyzed (Participants) | 36 | 33
  Change at week 4 | 0 [-10 to 10] | 10 [0 to 30]
Statistical Analysis 1: Comparison: Oral Iron vs Intravenous Iron; Between-group analysis of change at week 4; Test type: Other; p = 0.009, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was < 0.05

ADVERSE EVENTS:
Time Frame: Up to approximately 12 weeks
Description: Participants reported adverse events (AEs) by survey using the terms listed. The week 4 survey asked participants to report AEs occurring from weeks 1 to 4 (may have been up to week 6; primary outcome analysis period) and the week 8 survey asked participants to report AEs occurring from weeks 5 to 8 (may have been up to week 12; secondary outcome analysis period).
Groups:
- Oral Iron - Weeks 1 to 4: Adverse events occurring in the oral iron group during weeks 1 to 4
- Intravenous Iron - Weeks 1 to 4: Adverse events occurring in the intravenous iron group during weeks 1 to 4
- Oral Iron - Weeks 5 to 8: Adverse events occurring in the oral iron group during weeks 5 to 8
- Intravenous Iron - Weeks 5 to 8: Adverse events occurring in the intravenous iron group during weeks 5 to 8
Arm/Group | Oral Iron - Weeks 1 to 4 | Intravenous Iron - Weeks 1 to 4 | Oral Iron - Weeks 5 to 8 | Intravenous Iron - Weeks 5 to 8
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 17/40 | 15/40 | 13/40 | 9/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Iron - Weeks 1 to 4 (N=40) | Intravenous Iron - Weeks 1 to 4 (N=40) | Oral Iron - Weeks 5 to 8 (N=40) | Intravenous Iron - Weeks 5 to 8 (N=40)
Nausea/ Vomiting (Gastrointestinal disorders) | 8 | 7 | 3 | 2
Constipation (Gastrointestinal disorders) | 10 | 6 | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 2 | 2
Gastrointestinal symptoms not listed (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 1
Headache (Nervous system disorders) | 2 | 1 | 0 | 2
Edema/ Swelling of limbs (Blood and lymphatic system disorders) | 1 | 5 | 0 | 3
Itching (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 2
Body aches/ pains (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT04253626/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT04253626/ICF_000.pdf